CLINICAL TRIAL: NCT02456285
Title: Colorectal Cancer With Liver-limited Synchronous Metastases: an Inception Cohort Study of Standardised Care Pathways
Acronym: CoSMIC
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: University of Warwick (Other)
Responsible Party: Sponsor
Other Study IDs: R03880
Record Dates: First submitted 2015-05-20; First posted 2015-05-28 (Estimated); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Primary/Bowel-first Surgery — Patients undergoing primary/bowel-first surgery as part of a staged curative procedure. The liver metastases will be resected in a second planned operation.
Procedure: Liver-first surgery — Patients undergoing liver-first surgery as part of a staged curative procedure. The colorectal primary will be resected in a second planned operation.
Procedure: Synchronous resection surgery — Patients undergoing a synchronous colorectal primary resection and liver resection in a single operation.
Procedure: No surgery — Patients who have no surgery.

SUMMARY:
Background When first diagnosed, colorectal cancer has already metastasized in about 20% of patients to the liver or further (termed synchronous disease). For patients with metastatic disease limited to the liver, major surgery to resect both the primary colorectal cancer and the liver metastasis provides 5-year survival rates of 25-40%.

Conventional surgery removes the colorectal primary first, followed by adjuvant chemotherapy, and then resection of the liver metastasis. Surgical advances make synchronous resection (removing both primary and liver metastasis together) and liver-first resection possible.

Currently, there is no conclusive evidence to show which approach improves morbidity or survival, and therefore there is no optimum clinical pathway. Treatment is decided at multidisciplinary team (MDT) meetings and is dependent on multiple factors: cancer staging, patient health and preferences, and clinical experience.

Methods "Colorectal cancer with Synchronous liver-limited hepatic Metastasis: an Inception Cohort (CoSMIC)", will consent and recruit patients with a new diagnosis of synchronous colorectal cancer limited to the liver.

Patients will be recruited at Manchester Royal Infirmary (a National Health Service (NHS) regional cancer-network approved Hepato-pancreato-biliary specialist centers over 2 years using standardized data collection. The sequence of treatment received by each patient, and factors influencing treatment decisions, will be recorded and evaluated against European Society of Medical Oncology guidelines. The effect of surgery on patient quality of life, morbidity, mortality and the long-term outcome will be measured and compared for different treatment sequences adjusted for prognostic factors.

Anticipated Outputs and Value of Findings Direct comparison of conventional and new surgical sequences will be explored. Patient engagement, use of standardised recording, identifying common clinical patterns and decision making, and understanding sources of variation are essential steps to develop a definite randomized control trial to resolve the optimal clinical pathway.

DETAILED DESCRIPTION:
Patients who present with metastatic liver disease following treatment of the primary (termed metachronous disease) receive care focused on this new metastatic disease. In contrast, the management of patients who present with colorectal cancer and concurrent liver metastases (synchronous metastasis) is more complex. These patients may have less favourable cancer biology and thus may be less likely to become long-term survivors. Logically, the management of patients with colorectal cancer with synchronous metastases can be dichotomised into those with hepatic disease together with extra-hepatic metastatic disease and those with liver-limited metastatic disease. In the first category, systemic chemotherapy is the mainstay of treatment advocated in current guidelines for patients with advanced multi-site metastatic (liver and systemic metastatic) disease of colorectal cancer origin.

The second category of patients with liver-limited synchronous metastases represents a complex and common clinical management problem. Traditional management (referred to variously as the classical or staged approach) comprised resection of the colorectal primary tumour followed by adjuvant chemotherapy with liver resection being undertaken as a subsequent operation. Advances in surgery, anaesthesia and critical care have made two alternative options feasible for patients with synchronous disease. The first is synchronous resection of the liver metastases and the colorectal primary. This has the attraction of removing the macroscopic tumour burden with a single operation. However, the morbidity of complex liver resection combined with major bowel resection may be considerable and there is some evidence of a negative effect on progression-free survival. The second option in the management of synchronous disease is resection of the liver metastatic disease as the first step, termed the reverse or liver-first approach. Liver-first surgery to manage synchronous colorectal cancer and liver metastatic disease has become more widely utilised because of oncological and technical developments. Oncologically, evidence of improved outcome in locally advanced rectal cancer treated by pre-operative chemo-radiotherapy prior to surgical resection creates a potential "window" in which liver resection may be undertaken. The technical development of colonic stenting permits symptoms associated with rectal cancer such as partial obstruction to be palliated without recourse to urgent bowel surgery. The liver-first strategy may be oncologically advantageous if liver metastatic disease rather than the primary cancer gives rise to systemic metastasis - although this is not established. A further potentially important benefit of the liver-first approach is that pelvic surgery may be either avoided or less extensive in patients with rectal tumours with a complete endoscopic, radiological and clinical response to chemo-radiotherapy.

Currently, evidence is inadequate to inform the selection of treatment for patients with colorectal cancer with synchronous liver-limited hepatic metastases. Specifically, in these patients, optimal pathways are not defined and there is a dearth of prospectively recorded cohort- defining factors influencing treatment selection or outcome. Given the treatment permutations to be understood, an inception cohort study would allow us to understand patient outcomes as a function of clinical decisions and patient/disease characteristics. By limiting care available to patients to a common evidence-informed pathway, sources of treatment variation can be minimised and, within a prospective design, data quality be optimised with respect to patient and treatment characteristics.

Following informed consent and recruitment, data will be collected on patients with colorectal cancer with liver-limited hepatic metastases including patient variables, treatment selection, factors influencing treatment, treatment-related morbidity and outcome. Regression modelling of findings will permit influences of patient and treatment factors upon outcomes to be quantified. Patterns of clinical decision making will help to understand the characteristics of patients for whom equipoise exists or is absent.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Able to give informed consent
* Have a histological diagnosis of colorectal cancer
* No prior history of malignancy
* Have radiological evidence on either contrast-enhanced computed tomography or contrast-enhanced magnetic resonance scanning of hepatic metastases at the time of diagnosis of the primary tumour or within 3 months thereof. Liver metastases should not be biopsied.
* Computed tomographic and/or 18fluoro-deoxyglucose positron emission tomographic (FDG-PET) evidence of the absence of extrahepatic metastases.
* Magnetic resonance scan assessment of local stage of rectal primary tumours.
* World Health Organisation performance status (PS) 0, 1 or 2 and considered by multidisciplinary team to be suitable for chemotherapy.
* Consent to allow surplus pathological material to be analysed for translational research projects (patients may decline participation in this supplementary component and still participate in the main trial).

Exclusion Criteria:

* Patients who are under 18 years of age.
* Patients who are unable to give informed consent.
* Patients who are unfit for the chemotherapy regimens in this protocol.
* Any psychiatric or neurological condition assessed by clinical judgement to compromise the patient's ability to give informed consent or to comply with oral medication.
* Partial or complete bowel obstruction not amenable to resolution by stent or diversion.
* Pre-existing neuropathy (> grade 1).
* Patients with another previous or current malignant disease.
* Patients with known hypersensitivity reactions to any of the components of the study treatments.
* Patients with distant metastases outwith the liver.
* Patients who have received prior chemotherapy with oxaliplatin.
* Patients with a personal or family history suggestive of dihydropyrimidine dehydrogenase (DPD) deficiency or with known DPD deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients with colorectal cancer with liver-limited hepatic metastases referred to the Hepatobiliary Surgical Unit at Manchester Royal Infirmary - a National Health Service (NHS) regional cancer-network approved hepato-pancreato-biliary (HPB) centre with a formally constituted and National Cancer Network peer-review accredited multidisciplinary team (MDT).
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Adherence to an evidence-informed common pathway assessed using guidelines suggested by the European Society of Medical Oncology (ESMO) | 2 years
  The first primary outcome measure of CoSMIC is to assess the adherence to an evidence-informed common pathway, using guidelines suggested by the European Society of Medical Oncology (ESMO). These include early use of neo-adjuvant chemotherapy, surgical resection and adjuvant chemotherapy as the final stage. The treatment options within the common pathway standardise initial staging, accommodating treatment for liver metastases according to liver involvement and location of disease as well as different treatment requirements for patients with rectal primary cancer compared to those with colonic primary tumours.

CONTACTS AND LOCATIONS:
Overall Officials: Ajith K Siriwardena, MD, FRCS, Principal Investigator — Hepatobiliary Surgery Unit, Manchester Royal Infirmary, United Kingdom; James Mason, DPhil, Study Director — Durham Clinical Trials Unit, Wolfson Research Institute, Durham University, United Kingdom
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom

REFERENCES:
- [Background] Siriwardena AK, Mason JM, Mullamitha S, Hancock HC, Jegatheeswaran S. Management of colorectal cancer presenting with synchronous liver metastases. Nat Rev Clin Oncol. 2014 Aug;11(8):446-59. doi: 10.1038/nrclinonc.2014.90. Epub 2014 Jun 3. PMID 24889770
- [Background] Jegatheeswaran S, Mason JM, Hancock HC, Siriwardena AK. The liver-first approach to the management of colorectal cancer with synchronous hepatic metastases: a systematic review. JAMA Surg. 2013 Apr;148(4):385-91. doi: 10.1001/jamasurg.2013.1216. PMID 23715907
- [Derived] Chan AKC, Mason JM, Baltatzis M, Siriwardena AK; CoSMIC Collaborators. Management of Colorectal Cancer with Synchronous Liver Metastases: An Inception Cohort Study (CoSMIC). Ann Surg Oncol. 2022 Mar;29(3):1939-1951. doi: 10.1245/s10434-021-11017-7. Epub 2021 Oct 30. PMID 34716838
- [Derived] Siriwardena AK, Chan AKC, Ignatowicz AM, Mason JM; CoSMIC study collaborators. Colorectal cancer with Synchronous liver-limited Metastases: the protocol of an Inception Cohort study (CoSMIC). BMJ Open. 2017 Jun 9;7(6):e015018. doi: 10.1136/bmjopen-2016-015018. PMID 28601828